CLINICAL TRIAL: NCT01986036
Title: The Acute, Synergistic Effects of Protein and Calcium on Appetite and Energy Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD, Research Fellow, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 32AN4
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Proteins; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CONTROL (Sham Comparator): Control breakfast low in protein and calcium. Porridge-based breakfast.
  Interventions: Dietary Supplement: Porridge-based breakfast.
- PROTEIN (Active Comparator): High-protein breakfast.
  Interventions: Dietary Supplement: Protein; Dietary Supplement: Porridge-based breakfast.
- CALCIUM (Active Comparator): High-calcium breakfast.
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Porridge-based breakfast.
- PRO-CAL (Experimental): High-protein and calcium breakfast.
  Interventions: Dietary Supplement: Protein; Dietary Supplement: Calcium; Dietary Supplement: Porridge-based breakfast.

INTERVENTIONS:
Dietary Supplement: Protein — Milk-Protein
  Arms: PRO-CAL; PROTEIN
Dietary Supplement: Calcium — Soluble calcium powder.
  Arms: CALCIUM; PRO-CAL
Dietary Supplement: Porridge-based breakfast. — Oats and water.

SUMMARY:
High-protein meals have previously been shown to acutely reduce appetite and energy intake. More recently, meals higher in calcium have also been shown to increase feelings of fullness, circulating insulin and intestinal peptide concentrations and reduce appetite sensations.

This study aims to assess whether calcium and protein act synergistically to acutely influence appetite and energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* BMI 18.5-29.9 kg/m2
* Age: 18-40 years

Exclusion Criteria:

* Smokers
* Food allergies
* Metabolic disorders (ie. type 2 diabetes)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Energy Intake | 60 min post test-meal
  Energy intake will be assessed by ad libitum consumption of a homogenous pasta meal, 1 h after the test-meal.

SECONDARY OUTCOMES:
Subjective appetite sensations | 1 hr
  Subjective appetite sensations (hunger, satisfaction, prospective consumption and fullness) will be assessed by visual analogue scales at baseline, and every 15 min following test-meal consumption.
Insulin concentrations | 1 hr
  Plasma insulin concentrations will be determined at baseline and every 15 min following test-meal consumption.
GLP-1 (7-36) concentrations | 1 hr
  Plasma glucagon-like peptide-1 (GLP-1) (7-36) concentrations will be determined at baseline and every 15 min following consumption of the test meal.
GIP concentration | 1 hr
  Plasma glucose-dependent insulinotropic peptide (GIP) concentrations will be determined at baseline and evert 15 min following test-meal consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Javier T Gonzalez, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] Astbury NM, Stevenson EJ, Morris P, Taylor MA, Macdonald IA. Dose-response effect of a whey protein preload on within-day energy intake in lean subjects. Br J Nutr. 2010 Dec;104(12):1858-67. doi: 10.1017/S000711451000293X. Epub 2010 Sep 28. PMID 20875183
- [Background] Gonzalez JT, Rumbold PL, Stevenson EJ. Appetite sensations and substrate metabolism at rest, during exercise, and recovery: impact of a high-calcium meal. Appl Physiol Nutr Metab. 2013 Dec;38(12):1260-7. doi: 10.1139/apnm-2013-0056. Epub 2013 Jun 18. PMID 24195627
- [Background] Gonzalez JT, Stevenson EJ. Calcium co-ingestion augments postprandial glucose-dependent insulinotropic peptide(1-42), glucagon-like peptide-1 and insulin concentrations in humans. Eur J Nutr. 2014;53(2):375-85. doi: 10.1007/s00394-013-0532-8. Epub 2013 May 21. PMID 23689561
- [Derived] Gonzalez JT, Green BP, Brown MA, Rumbold PL, Turner LA, Stevenson EJ. Calcium ingestion suppresses appetite and produces acute overcompensation of energy intake independent of protein in healthy adults. J Nutr. 2015 Mar;145(3):476-82. doi: 10.3945/jn.114.205708. Epub 2015 Jan 14. PMID 25733462